CLINICAL TRIAL: NCT00760942
Title: Randomized Study of a Liquid High-Calorie Preterm Formula Versus Powdered Human Milk Fortifier in Very-Low Birthweight Infants
Brief Title: Liquid Preterm Formula Versus Powdered Human Milk Fortifier in VLBW Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14132
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Infant, Very Low Birth Weight
Keywords: Low birth weight; neonates; premature infants; nutrition; human milk fortification; Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Liquid human milk fortifier
  Interventions: Dietary Supplement: Similac special care 30
- 2 (Active Comparator): Powdered human milk fortifier
  Interventions: Dietary Supplement: Similac human milk fortifier

INTERVENTIONS:
Dietary Supplement: Similac special care 30 — Liquid pre-term formula 30Kcals/oz. used as human milk fortifier.
  Arms: 1
Dietary Supplement: Similac human milk fortifier — Powdered human milk fortifier.
  Arms: 2

SUMMARY:
This study aims to compare the short-term effects on growth and feeding tolerance of a liquid high calorie formula added to human milk versus powdered human milk fortifier in small preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 500 and 1499 grams of birthweight, receiving mother's milk.

Exclusion Criteria:

* Infants with major congenital anomalies and previous history of gastrointestinal disease.

Ages: 1 Day to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be weight gain in g/kg/d over the observation period. Body weight will be measured daily. | 2 - 6 weeks

SECONDARY OUTCOMES:
Hospital stay and feeding intolerance | 2-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Willeitner, M.D., Principal Investigator — University of Oklahoma
Locations (1):
- Neonatal Intensive Care Unit/Children's Hospital, Oklahoma City, Oklahoma, United States